CLINICAL TRIAL: NCT00760487
Title: Visual Function After Implantation of Bilateral AcrySof® Toric Natural Intraocular Lens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Ms Myrna Bergen, Phase IV Clinical Research Manager, Alcon Canada Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALCONsurtor001.06
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2010-04-07 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Cataract
Keywords: Cataract AcrySof Toric IOL; Bilateral cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AcrySof Toric IOL (Experimental): AcrySof Toric Intraocular Lens (IOL)
  Interventions: Device: AcrySof Toric IOL

INTERVENTIONS:
Device: AcrySof Toric IOL — Implantation with the AcrySof Toric IOL for cataract replacement and multiple follow-up assessments

SUMMARY:
The purpose of this study is to evaluate the effect that placement and power of the AcrySof Toric has on post-operative visual acuity and spectacle independence for distance vision. This will be determined by comparing manifest refraction pre-operatively and post-operatively and by evaluating the rotational stability of the lens over time.

ELIGIBILITY:
Inclusion Criteria:

* Are a candidate for bilateral implantation
* In good general and ocular health, 21 years of age or older, of either gender or any race, diagnosed with age-related cataracts in both eyes
* In need of spherical correction between 10.0 Diopter (D) and 30.0 D
* Preoperative regular corneal astigmatism, ≥ 1.0 D and ≤ 2.5 D , as measured by keratometry
* Willing and able to complete all required postoperative visits
* Able to comprehend and sign a statement of informed consent
* Pupil dilation ≥ 6.0 mm
* Expected to achieve a postoperative logMAR +0.3 or better visual acuity (as assessed by one or more of the following: fundus examination, pinhole visual acuity, and/or PAM evaluation);

Exclusion Criteria:

Exclusion Criteria Before Surgery - Ocular

* Previous cataract patient without potential of bilateral implantation
* Females of child bearing potential
* Irregular corneal astigmatism
* Keratopathy/Keratectasia - any corneal abnormality including but not limited to the following: keratoconus, keratoglobus, keratolysis, keratomalacia, keratomycosis, and cornea plana
* Any inflammation or edema (swelling) of the cornea, including but not limited to the following: keratitis, keratoconjunctivitis, and keratouveitis
* Previous corneal reshaping, including but not limited to the following: keratomileusis, radial keratotomy (RK), photorefractive keratectomy (PRK), Laser in Situ Keratomileusis (LASIK), Thermal Keratoplasty (TK), and Penetrating Keratoplasty (PK)
* Clinically significant corneal dystrophy (including Fuch's dystrophy)
* Previous corneal transplant
* Amblyopia
* Glaucoma (medically uncontrolled)
* Clinically significant RPE/Macular changes
* Proliferative diabetic retinopathy
* History of macular edema
* Previous history of retinal detachment
* History of uveitis/iritis
* Extremely shallow anterior chamber, not due to swollen cataract
* Iris neovascularization
* Microphthalmos
* Absent eye or eye with no light perception (NLP) as fellow eye
* Rubella, congenital, traumatic, or complicated cataract
* Optic atrophy

Exclusion Criteria During Surgery

* Other procedures at this surgery
* Limbal relaxing incisions (LRIs) or any other procedure to reduce the amount of preoperative astigmatism on the study eye(s), whether implanted with SA60TT or SA60AT, for the duration of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects >21 years of age, either sex and any race. Diagnosis of cataracts in one or both eyes.
Pre-assignment Details: Subject's eligibility was determined at the preoperative visit. All subjects met inclusion/exclusion criteria.
Groups:
- AcrySof Toric IOL: Implantation of the AcrySof Toric Intraocular lens (IOL)
Period: Overall Study
Arm/Group | AcrySof Toric IOL
Started | 120
Completed | 117
Not Completed | 3
Not completed — Unilateral implantation | 3

BASELINE CHARACTERISTICS:
Arm/Group | AcrySof Toric IOL
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 77
  >=65 years | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 41

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (VA)
Description: Pre-operative and 1 month, 3 month, and 6 month post-operative visual acuity (VA) measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". It is a unit of measure for visual acuity (VA).
Time Frame: Pre-operative, 1 month, 3 month, and 6 month post-operative
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | AcrySof Toric IOL
Number analyzed (Participants) | 117
logMAR
  Pre-Operative | 0.7 (0.06)
  1 Day Post-operative | 0.06 (0.12)
  3 Months Post-operative | 0.05 (0.11)
  6 Months Post-operative | 0.05 (0.11)

2. Secondary Outcome: Spectacle Independence
Description: Percentage of subjects reporting that they never wear glasses at the 6 month post-operative visit
Time Frame: 6 months post-operative
Measure: Number; unit: Percentage of participants
Arm/Group | AcrySof Toric IOL
Number analyzed (Participants) | 117
Percentage of participants | 69

3. Secondary Outcome: IOL Rotation
Description: Evaluation of percentage of patients that experienced rotation of the intraocular lens (IOL) less than or equal to 5 degrees from initial implantation, and less than or equal to 10 degrees from initial implantation.
Time Frame: 6 months post-operative
Measure: Number; unit: Percentage of Participants
Arm/Group | AcrySof Toric IOL
Number analyzed (Participants) | 117
Percentage of Participants
  Less than or equal to 5 degrees | 91
  Less than or equal to 10 degrees | 99

ADVERSE EVENTS:
Arm/Group | AcrySof Toric IOL
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 1/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AcrySof Toric IOL (N=120)
Lens Repositioning (Surgical and medical procedures) | 1 (1) — Repositioning of the intraocular lens during outpatient procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor Condfidential information will be submitted for publication without Sponsor's prior written agreement.